CLINICAL TRIAL: NCT05138731
Title: LC-MS Based Metabolomics Study of Coronary Heart Disease: Diagnostic and Prognostic Value of Metabolites
Brief Title: Metabolomics Profiling of Coronary Heart Disease
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: General Hospital of Ningxia Medical University (Other)
Responsible Party: Principal Investigator, Jun He, vice director of the department of cardiovascular internal medicine, General Hospital of Ningxia Medical University
Other Study IDs: JH
Record Dates: First submitted 2021-11-17; First posted 2021-12-01 (Actual); Last update posted 2022-01-14 (Actual); Status verified 2021-12

CONDITIONS: Biomarkers
Keywords: metabolomics; biomarkers; liquid chromatography-mass spectrometry; coronary artery disease; serum; urine
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum and urine samples from all participants
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (7):
- Stable angina (SA): Typical chronic exersive angina pectoris attacks, lasting several minutes to more than 10 minutes, 3-5 minutes in most cases, generally not more than 30 minutes. The pain disappeared after rest or taking nitrates, and the pain degree, frequency, duration, nature and inducing factors did not change in the last 1-3 months.
  Interventions: Other: treatments according guidelines
- Unstable angina (UA）: Including resting angina (attack at rest, the duration is usually >20 minutes), primary angina (usually the first symptoms within 1-2 months, very light physical activity can be induced, at least CCSIII level), worsening angina (angina gradually increases on the basis of relatively stable labor angina. More severe pain, longer or more frequent pain, at least grade I increase according to THE CCS classification, at least GRADE II CCSI). TNI was negative, routine electrocardiogram may have transient ST segment depression, T wave low flat or inverted.
  Interventions: Other: treatments according guidelines
- Acute non-ST-segment elevation myocardial infarction （NSTEMI）: Patients with elevated troponin accompanied by one or more of the following conditions: electrocardiogram showed new ST segment depression or T wave flatness or inversion; Persistent ischemic chest pain; Echocardiography showed abnormal segmental ventricular wall activity. Abnormal coronary angiography.
  Interventions: Other: treatments according guidelines
- Acute ST-segment elevation myocardial infarction （STEMI）: Troponin was elevated, and ECG showed ST segment arcuate back elevation, accompanied by one or more of the following conditions: persistent ischemic chest pain; Echocardiography showed segmental abnormal ventricular wall activity; Abnormal coronary angiography.
  Interventions: Other: treatments according guidelines
- normal coronary artery （NCA）: symptoms of chest pain and no stenosis in coronary arteries (such as myocardial bridging, reflux esophagitis, intercostals neuralgia, cervical spondylopathy, and unexplained chest pain)
  Interventions: Other: treatments according guidelines
- nonobstructive coronary atherosclerosis （NOCA）: stenosis < 50% in coronary arteries
  Interventions: Other: treatments according guidelines
- healthy volunteers: Healthy control subjects who had no significant systemic diseases (e.g. ischemic heart disease, hypertension,diabetes,cancer, pulmonary disease, or infectious diseases) were recruited from Physical Examination Center of Ningxia Medical University General Hospital

INTERVENTIONS:
Other: treatments according guidelines — different group intervened with different treatment following guidelines/consensuses accordingly
  Groups: Acute ST-segment elevation myocardial infarction （STEMI）; Acute non-ST-segment elevation myocardial infarction （NSTEMI）; Stable angina (SA); Unstable angina (UA）; nonobstructive coronary atherosclerosis （NOCA）; normal coronary artery （NCA）

SUMMARY:
This study sought to assess the diagnostic and prognostic values of metabolomics in coronary artery disease(CAD).

DETAILED DESCRIPTION:
The purpose of this study is to establish a powerful diagnostic and prognostic model based on metabolites in CAD patients.A total of 821 hospitalized patients with CAD and 200 healthy volunteers are enrolled.Specifically, 200 CAD patients from single-centre are regarded as discovery set, 300 CAD patients from multicentre are regarded as validation set. A third independent set including 321patitents is regarded as application set. Untargeted and targeted metabolomics analysis about serum and urine samples in all subjects will be performed using high-performance liquid chromatography coupled with mass spectrometry technology. Univariate and multivariate analysis methods are used to extract and analyze the differential mebabolites. By exploring the relationship between the differential mebabolites and clinical manifestions, a set of diagnostic biomarkers for CAD will be identified. By elucidating the correlation between the differential mebabolites and MACEs, a effective prognostic model will be established. Adverse events are defined as the combined endpoints of death or major adverse cardiovascular events(MACEs) in patients with CAD for at least 1 year follow-up after discharge. In brief, we aim to establish valuabe diagnostic and predictive models based on novel baseline metabolites in patients with CAD.

ELIGIBILITY:
Inclusion Criteria:

* Objective evidence of coronary heart disease risk factors
* Or angina pectoris symptoms
* Or ECG ischemic changes
* Or elevated myocardial enzymes, myocardial radionuclide scanning showing myocardial filling defect, coronary CT showing coronary stenosis ≥ 50%

Exclusion Criteria:

* Older than 80 years and younger than 18 years old,
* Aortic dissection
* Pulmonary embolism
* Malignant tumor
* Autoimmune diseases
* Systemic systemic diseases
* Severe infectious diseases
* Trauma, surgery in the last three months
* Myocarditis, cardiomyopathy, pericarditis, severe congenital heart disease
* Syphilis
* Human immunodeficiency virus / acquired immunodeficiency syndrome
* Hepatitis B and hepatitis C

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: About 821 subjects will be recruited from 5 centers in different hospitals.
Sampling Method: Probability Sample
Enrollment: 821 (Estimated)
Dates: Start 2020-10-01 (Actual); Primary Completion 2023-01-30 (Estimated); Study Completion 2023-05-30 (Estimated)

PRIMARY OUTCOMES:
Death | Follow-up is expected to end on December 30, 2022
  A composite of death from cardiovascular causes in patients with CAD

SECONDARY OUTCOMES:
Major adverse cardiovascular events | Follow-up is expected to end on December 30, 2022
  Hospitalization for recurrent severe angina pectoris, acute myocardial infarction, revascularization, malignant arrhythmia, new heart failure or acute attack of chronic heart failure, cardiac arrest and stroke.

CONTACTS AND LOCATIONS:
Overall Officials: Hechun Xia, MA, Study Chair — General Hospital of Ningxia Medical University
Locations (5):
- China (5):
  - Department of Cardiovascular Internal Disease, Guyuan People's Hospital of Ningxia Autonomous Region, Guyuan, Ningxia
  - Fifth People's Hospital of Ningxia Autonomous Region, Shizuishan, Ningxia
  - Affiliated Cardio-Cerebrovascular Hospital of Ningxia Medical University, Yinchuan, Ningxia
  - People's Hospital of Ningxia Hui Autonomous Region, Yinchuan, Ningxia
  - Department of Cardiaovascular Internal Disease, General Hospital of Ningxia Medical University, Yinchuan, Ningxia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Iida M, Harada S, Takebayashi T. Application of Metabolomics to Epidemiological Studies of Atherosclerosis and Cardiovascular Disease. J Atheroscler Thromb. 2019 Sep 1;26(9):747-757. doi: 10.5551/jat.RV17036. Epub 2019 Aug 2. PMID 31378756
- [Background] Vaarhorst AA, Verhoeven A, Weller CM, Bohringer S, Goraler S, Meissner A, Deelder AM, Henneman P, Gorgels AP, van den Brandt PA, Schouten LJ, van Greevenbroek MM, Merry AH, Verschuren WM, van den Maagdenberg AM, van Dijk KW, Isaacs A, Boomsma D, Oostra BA, van Duijn CM, Jukema JW, Boer JM, Feskens E, Heijmans BT, Slagboom PE. A metabolomic profile is associated with the risk of incident coronary heart disease. Am Heart J. 2014 Jul;168(1):45-52.e7. doi: 10.1016/j.ahj.2014.01.019. Epub 2014 Apr 4. PMID 24952859
- [Background] Cavus E, Karakas M, Ojeda FM, Kontto J, Veronesi G, Ferrario MM, Linneberg A, Jorgensen T, Meisinger C, Thorand B, Iacoviello L, Bornigen D, Woodward M, Schnabel R, Costanzo S, Tunstall-Pedoe H, Koenig W, Kuulasmaa K, Salomaa V, Blankenberg S, Zeller T; BiomarCaRE consortium. Association of Circulating Metabolites With Risk of Coronary Heart Disease in a European Population: Results From the Biomarkers for Cardiovascular Risk Assessment in Europe (BiomarCaRE) Consortium. JAMA Cardiol. 2019 Dec 1;4(12):1270-1279. doi: 10.1001/jamacardio.2019.4130. PMID 31664431
- [Background] McGarrah RW, Crown SB, Zhang GF, Shah SH, Newgard CB. Cardiovascular Metabolomics. Circ Res. 2018 Apr 27;122(9):1238-1258. doi: 10.1161/CIRCRESAHA.117.311002. PMID 29700070
- [Background] Fan Y, Li Y, Chen Y, Zhao YJ, Liu LW, Li J, Wang SL, Alolga RN, Yin Y, Wang XM, Zhao DS, Shen JH, Meng FQ, Zhou X, Xu H, He GP, Lai MD, Li P, Zhu W, Qi LW. Comprehensive Metabolomic Characterization of Coronary Artery Diseases. J Am Coll Cardiol. 2016 Sep 20;68(12):1281-93. doi: 10.1016/j.jacc.2016.06.044. PMID 27634119
- [Background] Hilvo M, Meikle PJ, Pedersen ER, Tell GS, Dhar I, Brenner H, Schottker B, Laaperi M, Kauhanen D, Koistinen KM, Jylha A, Huynh K, Mellett NA, Tonkin AM, Sullivan DR, Simes J, Nestel P, Koenig W, Rothenbacher D, Nygard O, Laaksonen R. Development and validation of a ceramide- and phospholipid-based cardiovascular risk estimation score for coronary artery disease patients. Eur Heart J. 2020 Jan 14;41(3):371-380. doi: 10.1093/eurheartj/ehz387. PMID 31209498
- [Background] Qin M, Zhu Q, Lai W, Ma Q, Liu C, Chen X, Zhang Y, Wang Z, Chen H, Yan H, Lei H, Zhang S, Dong X, Wang H, Huang M, Lian Q, Zhong S. Insights into the prognosis of lipidomic dysregulation for death risk in patients with coronary artery disease. Clin Transl Med. 2020 Sep;10(5):e189. doi: 10.1002/ctm2.189. PMID 32997403
- [Background] Zhang L, Wei TT, Li Y, Li J, Fan Y, Huang FQ, Cai YY, Ma G, Liu JF, Chen QQ, Wang SL, Li H, Alolga RN, Liu B, Zhao DS, Shen JH, Wang XM, Zhu W, Li P, Qi LW. Functional Metabolomics Characterizes a Key Role for N-Acetylneuraminic Acid in Coronary Artery Diseases. Circulation. 2018 Mar 27;137(13):1374-1390. doi: 10.1161/CIRCULATIONAHA.117.031139. Epub 2017 Dec 6. PMID 29212895
- See also: Application of Metabolomics to Epidemiological Studies of Atherosclerosis and Cardiovascular Disease — http://doi.org/10.5551/jat.RV17036
- See also: A metabolomic profile is associated with the risk of incident coronary heart disease — http://hub.pubmedplus.com/10.1016/j.ahj.2014.01.019
- See also: Association of Circulating Metabolites With Risk of Coronary Heart Disease in a European Population Results From the Biomarkers for Cardiovascular Risk Assessment in Europe (BiomarCaRE) Consortium — http://hub.pubmedplus.com/10.1001/jamacardio.2019.4130
- See also: Cardiovascular Metabolomics — http://hub.pubmedplus.com/10.1161/circresaha.117.311002
- See also: ComprehensiveMetabolomicCharacterization of Coronary Artery Diseases — http://dx.doi.org/10.1016/j.jacc.2016.06.044
- See also: Development and validation of a ceramide- and phospholipid-based cardiovascular risk estimation score for coronary artery disease patients — http://hub.pubmedplus.com/10.1093/eurheartj/ehz387
- See also: Insights into the prognosis of lipidomic dysregulation for death risk in patients with coronary artery disease. — http://hub.pubmedplus.com/10.1002/ctm2.189
- See also: Functional Metabolomics Characterizes a Key Role for N-Acetylneuraminic Acid in Coronary Artery Diseases — http://hub.pubmedplus.com/10.1161/circulationaha.117.031139